CLINICAL TRIAL: NCT04806581
Title: Clinical Study of Congener Allogeneic Hepatocyte Transplantation Treatment in Patients With Liver Cirrhosis
Brief Title: Clinical Study of Hepatocyte Transplantation for Liver Cirrhosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI-IM-001
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; allogeneic hepatocyte; transplantation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allogeneic Hepatocyte Cohort 1 (Experimental): Participants will each be administered L dose for one time. With 28days follow-up after the cells infusion.
  Allogeneic hepatocyte cell numbers: L
  Interventions: Drug: Allogeneic Hepatocyte
- Allogeneic Hepatocyte Cohort 2 (Experimental): Participants will each be administered M dose for one time. With 28days follow-up after the cells infusion.
  Allogeneic hepatocyte cell numbers: M
  Interventions: Drug: Allogeneic Hepatocyte
- Allogeneic Hepatocyte Cohort 3 (Experimental): Participants will each be administered H dose for one time. With 28days follow-up after the cells infusion.
  Allogeneic hepatocyte cell numbers: H
  Interventions: Drug: Allogeneic Hepatocyte

INTERVENTIONS:
Drug: Allogeneic Hepatocyte — Allogeneic hepatocyte with cell numbers L,M,H respectively.

SUMMARY:
The Primary Objective: To observe and determine the safety and tolerance of allogeneic hepatocyte transplantation in patients with liver cirrhosis and to establish the maximum-tolerated dose (MTD) and evaluate the dose-limiting toxicities (DLTs).

The Secondary Objective: To observe the therapeutic efficacy of allogeneic hepatocyte transplantation for liver cirrhosis.

DETAILED DESCRIPTION:
* A traditional 3 + 3 dose escalation design will be implemented.
* Successive cohorts of participants (3 or 3+3 participants /cohort) will start on a fixed cell numbers of allogeneic hepatocyte in three cohorts separately: L dose (low cell numbers); M dose (medium cell numbers); H dose (high cell numbers).
* The 1st cohort will be given dose of L.
* The 2nd cohort will be given dose of M.
* The 3rd cohort will be given dose of H.
* Dose escalation will continue until the maximum-tolerated dose (MTD). If no DLTs are observed for 28days after administration of the last dose, a new cohort will be enrolled at the next planned dose level. If DLTs are observed in 2 of the three participants, the MTD will be determined to be the dose administered to the previous cohort. If DLTs are observed in one participant in the cohort, another three participants will be treated with the same dose level. If the new three participants aren't observed DLTs, another cohort will be enrolled at the upper dose. If at least one of the new three ones are observed DLTs, the below dose will be the MTD.
* MTD will stopped by testing increasing up to the H dose.
* Toxicities will be graded using the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0).

ELIGIBILITY:
Key Inclusion Criteria:

* The age at the time of signing the informed consent from 18 to 70 years old (including the boundary value), both male and female;
* Clinical diagnosis of liver cirrhosis;
* Be able to understand and sign informed consent.

Key Exclusion Criteria:

* Combined with liver cancer or other malignant tumors;
* Patients who can't cooperate;
* Prothrombin time (PT) exceeded the upper limit of normal control for 3-5 seconds or more;
* International normalized ratio (INR) >1.5;
* PLT<60×109/L；
* Recently use of anticoagulant or antiplatelet drugs (last 7 days);
* Recently (last 4 weeks) had upper gastrointestinal bleeding or spontaneous celiac inflammation;
* Moderate or large amount of ascites;
* The investigator assesses that the patient is unable or unwilling to comply with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28days
  Observe the safety and tolerance after single infusion of hepatocyte.
Dose-Limiting Toxicities | 28days
  Observe the safety and tolerance after single infusion of hepatocyte.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, Doctor, Principal Investigator — Department of Liver Surgery, Renji Hospital affiliated to Shanghai Jiao Tong University
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No